CLINICAL TRIAL: NCT00215007
Title: Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial With Levofloxacin as Prophylaxis for Bacterial Infections in Immunocompromised Patients After Allogeneic Transplantation of Hematopoietic Stem Cells
Brief Title: Trial of Levofloxacin as Prophylaxis After Allogeneic Stem Cell Transplantation (SCT)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Levosta-CBF-02/04
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2004-02

CONDITIONS: Malignancy; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Neoplasms | interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin

SUMMARY:
The purpose of this study is to evaluate the efficacy of levofloxacin to prevent bacterial infections in the postneutropenic period in patients who have undergone allogeneic stem cell transplantation (SCT).

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic SCT
* Postneutropenic period
* Written consent

Exclusion Criteria:

* Fever
* Antibiotic therapy
* Neutropenia
* Refusal by the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Igor Wolfgang Blau, Dr., Study Chair — Charite, CBF, Berlin, Germany
Locations (1):
- Charite, CBF, Berlin, State of Berlin, Germany